CLINICAL TRIAL: NCT01966341
Title: A Randomized Controlled Trial Comparing a Collaborative Cognitive Behavioral Therapy / Hypnotherapy Program to Standard Medical Management in the Treatment of Pediatric Functional Gastrointestinal Disease
Brief Title: Collaborative Cognitive Behavioral Therapy / Hypnotherapy for Treatment of Pediatric Functional Gastrointestinal Disease
Acronym: CAPP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruiting or enrolling participants has halted prematurely and will not resume
Sponsor: Seton Healthcare Family (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR-13-108
Record Dates: First submitted 2013-09-19; First posted 2013-10-21 (Estimated); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Irritable Bowel Syndrome (IBS)
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Hypnosis; Parasympatholytics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine Management (Active Comparator): All patients will be given a prescription for the use of antispasmodics. If patients demonstrate symptoms consistent with constipation predominant IBS they will be treated with laxatives. If symptoms are more consistent with diarrhea predominant IBS they will be treated with bulking agents (fiber) +/- antibiotics. Patient will be called every week while enrolled in the study in order to titrate doses, and answer questions.
  Interventions: Drug: Routine Management
- CBT/ Hypnotherapy (Experimental): The CBT (cognitive behavior therapy) program will consist of 7 sessions that will encompass the following skills of Symptom monitoring, Stress Management, Coping Skills, Relaxation training, Problem solving, and Cognitive Restructuring.The hypnotherapy program will be modeled after the North Carolina Standardized Hypnosis Treatment for Irritable Bowel Syndrome
  Interventions: Behavioral: CBT/ Hypnotherapy

INTERVENTIONS:
Behavioral: CBT/ Hypnotherapy — The CBT program will consist of 7 sessions that will encompass the following skills of Symptom monitoring, Stress Management, Coping Skills, Relaxation training, Problem solving, and Cognitive Restructuring.The hypnotherapy program will be modeled after the North Carolina Standardized Hypnosis Treatment for Irritable Bowel Syndrome
  Arms: CBT/ Hypnotherapy
Drug: Routine Management — Treatment with use of antispasmodics,laxatives, and/or bulking agents (fiber) +/- antibiotics.
  Other Names: antispasmodics,laxatives,fiber,antibiotics.
  Arms: Routine Management

SUMMARY:
This program has been created to help patients with irritable bowel syndrome manage their symptoms and increase their functioning by using cognitive therapy skills and hypnosis.

DETAILED DESCRIPTION:
Functional Gastrointestinal Diseases (FGID) are a family disorders that are characterized by gastrointestinal symptoms in the absence of readily identifiable organic pathology. Examples of FGID include irritable bowel syndrome, rumination syndrome, and function constipation. These disorders are classically thought to stem from dysfunction of the enteric nervous system. However, there is a growing recognition that multiple factors play a role in the genesis of FGIDs. This idea is encapsulated by the "biopsychosocial" model of disease, and is supported by a body of literature which has identified higher rates of FGID in patients with anxiety, depression, post-traumatic stress disorder, agoraphobia, and other psychosocial dysfunction.

Recurrent Abdominal Pain and Irritable Bowel Syndrome are major causes of pediatric morbidity. Over a third of children and adolescents report recurrent abdominal pain, and the overall prevalence of non-organic abdominal pain has been noted to be over 75% 1 2. A large subset of these children report symptoms that are consistent with irritable bowel syndrome. Management of these children is complex and includes medical, dietary, and behavioral interventions. Medical therapy often revolves around the use of antispasmodics, probiotics, and antidepressants. The data supporting their use, however has been mixed.

Over the last twenty years behavioral therapies such as cognitive behavioral therapy (CBT) and hypnotherapy (HT) have come to light as major treatment modalities for functional gastrointestinal disease. In a large multicenter randomized controlled trial Levy et al compared 3-session CBT to a control intervention and noted significant improvements and pain and function in children 3. Similar results have been published in multiple smaller trials 4-8. Likewise, Vlieger et al compared hypnotherapy to standard medical therapy in 53 children with irritable bowel syndrome. They found that, while both interventions resulted in improved pain scores, the hypnotherapy group demonstrated lasting clinical improvement at 1 year followup 9. Five year follow-up data has recently been published and revealed that significantly more of the hypnotherapy group remained in remission without any further intervention 10. A growing body of literature is available validating the use of hypnotherapy in irritable bowel syndrome in adults, and pain syndromes more generally 11-14.

These therapies can be viewed as complementary to one another. CBT involves a very deliberate conscious understanding of ones disease process and triggers and focuses on successful pain mitigation measures. HT recruits the imagination with utilization of therapeutic imagery to down regulate inappropriate pain responses. Our center has developed a collaborative approach, utilizing both CBT and HT for the treatment of refractory IBS. To our knowledge no work has been done assessing the efficacy of such a collaborative approach using both CBT and HT in children with functional gastrointestinal disease. We therefore propose the following randomized case-control crossover trial to assess the efficacy our combined program.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 - 18
* Meets Rome III Criteria for Pediatric Irritable Bowel Syndrome

  * Abdominal discomfort or pain associated with 2 or more of the following at least 25% of the time
  * Improved with defecation
  * Onset associated with a change in frequency of stool
  * Onset associated with a change in form of the stool
  * No evidence of inflammatory, anatomic, metabolic, or neoplastic process that explains the subject's symptoms
  * Criteria fulfilled once per week for at least 2 months before diagnosis

Exclusion Criteria: Unwillingness / Inability to engage in cognitive behavioral therapy arm of study (weekly encounters with psychologist)

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Functional Disability Inventory (FDI) | 10 weeks
  The FDI is a measure of the degree to which children experience difficulty in physical and psychosocial functioning due to their physical health status. Respondents are asked to rate how much physical difficulty was perceived for a variety of everyday activities. Both child-report and parent-report versions are composed of 15 questions.

SECONDARY OUTCOMES:
Pain Beliefs Questionnaire | 10 weeks
  The Pain Beliefs Questionnaire is a 32-item measure assessing characteristic appraisals of pediatric abdominal pain severity (primary coping appraisals) and characteristic appraisals of ability to cope with pediatric abdominal pain (secondary coping appraisals).

OTHER OUTCOMES:
Pain Response Inventory (PRI) | 10 weeks
  The Pain Response Inventory (PRI) was developed as a multidimensional instrument to assess children's coping responses to recurrent pain
Pain Frequency Score / Pain Intensity Score (PFS/PIS) | 10 weeks
  Our primary outcome measure will be the PFS/PIS. It involves an aggregate score of pain intensity and frequency
Abdominal Pain Index (API; Walker, Smith, Garber, & Van Slyke, 1997) | 10 weeks
  Abdominal Pain Index comprises five items assessing the frequency, duration, and intensity of abdominal pain episodes experienced during the previous 2 weeks
Children's Somatization Inventory (CSI) | 10 weeks
  The CSI assesses a variety of nonspecific somatic symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Anees Siddiqui, MD, Principal Investigator — 'Specially for Children, Dell Children's Medical Center of Central Texas
Locations (1):
- 'Specially for Children, Dell Children's Medical Center of Central Texas, Austin, Texas, United States